CLINICAL TRIAL: NCT06008600
Title: KINO-DYSPNEA: Validation of Kinocardiography to Distinguish Dyspnea of Cardiac Origin From Others
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Tivoli (Other)
Collaborators: HeartKinetics (Unknown)
Responsible Party: Sponsor
Other Study IDs: P2021/414 / B4062021000223
Record Dates: First submitted 2023-05-30; First posted 2023-08-23 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Kinocardiography — Smartphone (application with seismocardiography)
  Other Names: NT-pro BNP blood measurement

SUMMARY:
Seismocardiography (SCG) measures the thoracic vibrations caused by the cardiac contraction and ejection of blood into the great vessels. Current smartphones with gyroscopes and accelerometers can measure these vibrations. Based on these components we measure and quantify the cardiac kinetic energy (kinocardiography) in order to differentiate dyspnea of cardiac origin from dyspnea of other origin. The study is conducted in an emergency service where a smartphone performs the measurement during 3 minutes. The results of the kinocardiography-based classification are then compared to the final diagnosis made by a physician. Currently, 235 patients have been included in the clinical study since May 2022. This rapid and non-invasive measurement allows the aid-to-diagnosis of heart failure without being influenced by other factors like the renal function for example that can be NT-pro BNP blood marker.

ELIGIBILITY:
Inclusion Criteria:

* Dyspnea.
* Adults aged above 18 years old.

Exclusion Criteria:

* Patients younger than 18 years old.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any adult presenting with dyspnea to the emergency department or cardiology consultation.
Sampling Method: Probability Sample
Enrollment: 528 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the ability of the Kinocardiography technique to discriminate cardiac caused dyspnea from others. | 18 months
  Area under the receiver operating characteristic curve (AUROC), negative predictive value (NPV) and specificity, with two-sided 95% CIs.

SECONDARY OUTCOMES:
Open retrospective exploratory study to validate the physiological interpretation of Kinocardiography in a clinical environment. | 18 months
  Establish a link between cardiac kinetic energy distribution in the cardiac cycle between major active clinical syndromes that may be concomitant in the field of cardiac disorders (hypertension, atrial fibrillation, ischemia, valvulopathy, heart-failure,…) and pulmonary (asthma, infection,..). These clinical diagnoses are supported by the physical examination and the patient's medical record at inclusion, with the aid of a measurement of troponin and NTBNP

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Tivoli, La Louvière, Hainaut, Belgium

REFERENCES:
- [Background] Hossein A, Rabineau J, Gorlier D, Pinki F, van de Borne P, Nonclercq A, Migeotte PF. Effects of acquisition device, sampling rate, and record length on kinocardiography during position-induced haemodynamic changes. Biomed Eng Online. 2021 Jan 6;20(1):3. doi: 10.1186/s12938-020-00837-5. PMID 33407507
- [Background] Morra S, Hossein A, Rabineau J, Gorlier D, Racape J, Migeotte PF, van de Borne P. Assessment of left ventricular twist by 3D ballistocardiography and seismocardiography compared with 2D STI echocardiography in a context of enhanced inotropism in healthy subjects. Sci Rep. 2021 Jan 12;11(1):683. doi: 10.1038/s41598-020-79933-4. PMID 33436841
- [Background] Morra S, Pitisci L, Su F, Hossein A, Rabineau J, Racape J, Gorlier D, Herpain A, Migeotte PF, Creteur J, van de Borne P. Quantification of Cardiac Kinetic Energy and Its Changes During Transmural Myocardial Infarction Assessed by Multi-Dimensional Seismocardiography. Front Cardiovasc Med. 2021 Mar 8;8:603319. doi: 10.3389/fcvm.2021.603319. eCollection 2021. PMID 33763456
- [Background] Hossein A, Rabineau J, Gorlier D, Del Rio JIJ, van de Borne P, Migeotte PF, Nonclercq A. Kinocardiography Derived from Ballistocardiography and Seismocardiography Shows High Repeatability in Healthy Subjects. Sensors (Basel). 2021 Jan 26;21(3):815. doi: 10.3390/s21030815. PMID 33530417